CLINICAL TRIAL: NCT02865915
Title: A Double-blind, Randomized, Parallel-group, Placebo-controlled Study of MLE4901 for the Treatment of Polycystic Ovary Syndrome (PCOS)
Brief Title: MLE4901 vs. Placebo for the Treatment of PCOS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The risk/benefit profile no longer indicated continued development.
Sponsor: Millendo Therapeutics US, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry); Covance (Industry)
Responsible Party: Sponsor
Organization: Millendo Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLE4901-101; 2016-002179-91 (EudraCT Number)
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: Acne; Hirsutism; Menstrual Irregularity; Alopecia
MeSH Terms: conditions — Polycystic Ovary Syndrome; Acne Vulgaris; Hirsutism; Menstruation Disturbances; Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Plain, round, biconvex, white film-coated tablets that appear identical to MLE4901 tablets
  Interventions: Drug: Placebo
- MLE4901 (Experimental): Plain, round, biconvex, white film-coated tablets administered twice per day
  Interventions: Drug: MLE4901

INTERVENTIONS:
Drug: MLE4901 — For 80% of subjects randomized to MLE4901 (n=24/30), the dose is 40 mg twice daily. Six subjects (20%) randomized to higher MLE4901 dose cohorts that were promptly discontinued.
  Arms: MLE4901
Drug: Placebo — Placebo to match active drug
  Arms: Placebo

SUMMARY:
This is a Phase 2b double-blind, randomized, parallel-group, placebo-controlled study of MLE4901 versus placebo in women with PCOS.

DETAILED DESCRIPTION:
Following a Screening/Wash-out Period of up to 12 weeks, an 8-week Lead-in Period (starting with a progestin challenge) will be used to better characterize the study population. A Treatment Period of 28 weeks' duration will follow the Lead-in Period. Then, an 8-week Follow-up Period (i.e., no study drug) will be used to assess the durability of effects of MLE4901. The study duration will be approximately 48 weeks (11 months) per subject

ELIGIBILITY:
Inclusion Criteria:

1. Oligo-/amenorrhea
2. At least one of the following during Screening:

   * Clinical signs of hyperandrogenism, where clinical hyperandrogenism may include hirsutism (defined as excessive terminal hair that appears in a male pattern), acne, or androgenic alopecia
   * Biochemical hyperandrogenism refers to an elevated serum androgen level (i.e., total, bioavailable or free testosterone level ≥ULN)
   * Polycystic ovarian morphology, defined as the presence of 12 or more follicles 2-9 mm in diameter and/or an increased ovarian volume >10 mL (without a cyst or dominant follicle) in either ovary
3. Body mass index (BMI) 22 to 45 kg/m2, inclusive
4. Must be willing to avoid use of all hair removal procedures and products during study participation
5. Must be willing to avoid all prescription treatments for acne and not increase the dose or frequency of their current non-prescription acne treatment regimen during study participation
6. Must be willing to avoid the use of all hair growth procedures and products during study participation
7. Permanently surgically sterilized (bilateral salpingectomy or tubal occlusion) >2 years or male partner(s) has had a vasectomy >2 years or must consent to use two permitted medically-acceptable methods of contraception throughout the study during any sexual intercourse with a male partner. Permitted medically-acceptable methods of birth control for this study are defined as use of a male condom plus one of the following: spermicide, diaphragm with spermicide, or an intrauterine device that does not contain steroid hormones.

Exclusion Criteria:

1. Menopausal or peri-menopausal, defined for this study as FSH (follicle stimulating hormone ) >10 IU/L
2. Irregular vaginal/menstrual bleeding caused by conditions other than PCOS (e.g., uterine polyps or submucosal uterine fibroids)
3. Abnormal Papanicolaou (Pap) test during Screening requiring follow-up sooner than 1 year after the test
4. Uncontrolled hypo- or hyperthyroidism
5. Post-hysterectomy or endometrial ablation
6. Post-oophorectomy (unilateral or bilateral) or other ovarian surgery
7. Medical history of type 1 or type 2 diabetes mellitus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Hope Research Institute, LLC, Phoenix, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Excell Research, Oceanside, California
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Avail Clinical Research, LLC, DeLand, Florida
  - Health Care Family Rehab & Research Center, Hialeah, Florida
  - University of Florida (UF), Jacksonville, Florida
  - Palmetto Professional Research, Miami, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Atlanta Women's Research Institute, Atlanta, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Womens Health Practice, Champaign, Illinois
  - GTC Enterprises LLC, Shawnee Mission, Kansas
  - Montana Health Research Institute, Inc., Billings, Montana
  - Upstate Clinical Research Associates, Williamsville, New York
  - PMG Research of Cary, Cary, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - University Hospitals Cleveland Medical Center, Mayfield Heights, Ohio
  - Clinical Research of Tiffin, Tiffin, Ohio
  - Main Line Fertility and Reproductive Medicine, Bryn Mawr, Pennsylvania
  - The Pennsylvania State University (Penn State) Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Perelman Center for Advanced Medicine - Penn Fertility Care, Philadelphia, Pennsylvania
  - Magnolia OB/GYN Research Center, Myrtle Beach, South Carolina
  - Texas Diabetes and Endocrinology, P.A. - South Austin, Austin, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Tidewater Clinical Research, Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 30 US sites. The study was initiated on 27 July 2016 and completed on 04 August 2017. Study sites consisted of a combination of private clinical research centers, medical clinics, and academic practices.
Pre-assignment Details: Prior to randomization, subjects completed a screening period with a wash-out of medications for PCOS symptoms (if needed). Eligible subjects then completed an 8-week Lead-in Period with an initial 5-day progestin challenge, self-report of menstrual bleeding, and assessment of ovulation status by urine pregnenediol-3-glucuronide.
Groups:
- Placebo Treatment Arm: Treatment with 1 matching placebo tablet self-administered twice daily
- MLE4901 Treatment Arm: Treatment with 1 tablet of MLE4901 self-administered twice daily [80% treated with dose of 40 mg twice daily]
Period: Overall Study
Arm/Group | Placebo Treatment Arm | MLE4901 Treatment Arm
Started | 25 | 30
Completed | 0 (Study terminated prior to completion by any subject) | 0 (Study terminated prior to completion by any subject)
Not Completed | 25 | 30
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Study terminated by sponsor | 23 | 18
Not completed — Dosing group discontinued | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo Treatment Arm: Matching placebo tablet self-administered twice daily
- Total: Total of all reporting groups
Arm/Group | Placebo Treatment Arm | MLE4901 Treatment Arm | Total
Number analyzed (Participants) | 25 | 30 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 30 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (5.16) | 28.5 (5.71) | 29.1 (5.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 22 | 27 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 20 | 24 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 30 | 55
Menstrual cycle frequency [Mean (Standard Deviation); unit: cycles/year] | 3.1 (1.74) | 2.8 (1.83) | 2.9 (1.78)

OUTCOME MEASURES:

1. Primary Outcome: Menstrual Cycle Duration
Description: Assessment of the number of days between menstrual cycles (i.e., days between the start of a menstrual period and the start of the next consecutive menstrual period) from baseline to end of 28 week double blind treatment period
Time Frame: 28 Week double blind treatment period
Population: The trial was terminated prior to collection of any efficacy data.
Groups:
- MLE4901 Treatment Arm: Treatment with 1 tablet of study drug self-administered twice daily (most dosed with 40 mg BID)
Arm/Group | Placebo Treatment Arm | MLE4901 Treatment Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Menstrual Periods
Description: Number of menstrual periods from baseline to the end of the 28 week double blind treatment period
Time Frame: 28 Week double blind treatment period
Population: Study terminated prior to collection of efficacy data.
Arm/Group | Placebo Treatment Arm | MLE4901 Treatment Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: During the time period between enrollment of the first subject until the data lock date, approximately 9 months.
Arm/Group | Placebo Treatment Arm | MLE4901 Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/30
Other Adverse Events (participants affected / at risk) | 15/25 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment Arm (N=25) | MLE4901 Treatment Arm (N=30)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment Arm (N=25) | MLE4901 Treatment Arm (N=30)
Nausea (Gastrointestinal disorders) | 5 (6) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Upper respiratory infection (Infections and infestations) | 5 (6) | 4 (4)
Streptococcal pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to termination of the study by the Sponsor, no patients completed the study. No efficacy data are available because study termination occurred prior to scheduled assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT02865915/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT02865915/SAP_001.pdf